CLINICAL TRIAL: NCT05398380
Title: Clinical Impact of Molecular Biomarkers in Liver Transplantation for Non-resectable Colorectal Liver Metastases: Translational Research
Brief Title: Liver Transplantation for Non-resectable Colorectal Liver Metastases: Translational Research
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Vall d'Hebron (Other)
Responsible Party: Principal Investigator, Cristina Dopazo Taboada, Consultant surgeon, MD/PhD, Hospital Vall d'Hebron
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METLIVER Study
Record Dates: First submitted 2022-05-20; First posted 2022-06-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-10

CONDITIONS: Colorectal Cancer; Liver Metastases; Genetic Change
Keywords: Liver Transplantation; Non-resectable colorectal liver metastases; Tumoral biomarkers; Translational research
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Liver Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transplantation (Experimental): Liver transplantation for the treatment of unresectable colorectal cancer liver metastases
  Interventions: Other: Liver transplantation

INTERVENTIONS:
Other: Liver transplantation — Liver transplantation

SUMMARY:
The patients with non-resectable colorectal liver metastases (CRLM) have always being considered a particular subgroup of CRLM in which the therapeutic approach, is focused on strategies that allow a potential surgery like neoadjuvant systemic treatments. But, the underlying biology that causes this particular profile of spread in a proportion of patients that always recur and progress in the liver has not been properly characterized from a biological point of view. Unfortunately, these patients finally develop liver metastasis not amenable for local treatments and become refractory to systemic treatments even without developing extrahepatic liver metastases. As a result, liver transplantation (LT) is a potential for patients without extrahepatic involvement and nonresectable CRLM. There are several studies that aims to evaluate if LT increases overall survival compared to best alternative care. To our knowledge, none of these studies incorporate objectives focused on the underlying tumor biology of this particular population and the development of focused strategies including a dynamic disease monitoring and targeted treatments for this particular population.The METLIVER trial will permit to expand the genetic studies to the whole complexity of metastatic lesions and a more precise evaluation of their genetic heterogeneity. Moreover, it will help to precise the type of genetic analyses on liquid biopsies that can be designed for patients that will unfortunately relapse mostly with lung metastases after LT. Our proposal will maximize the opportunity to produce an unprecedented knowledge on CRLM evolution and will provide new opportunities for relapsed patients.

DETAILED DESCRIPTION:
A prospective multicenter Spanish clinical phase II trial is proposed. The study population will consist of male and female with non-resectable CRLM, who are 18 to 70 years old, inclusive, at the time of providing informed consent. Patients will be identified, treated and followed by the clinical investigators within the different centers included in the present study. Those patients deemed unresectable CRLM by consensus in multidisciplinary meeting will be pre-screened for eligibility to be included in the study. After receiving the corresponding chemotherapy and if the patient meets the inclusion criteria and none of the exclusion criteria will sign the informed consent and will be evaluated for liver transplantation according to institutional protocols at the transplant unit. Patients eligible for liver transplantation will continue chemotherapy until the time of an organ is available. However, patients receiving treatment with bevacizumab or aflibercept will discontinue this treatment at time of inclusion in waiting list. If there are no further contraindications at the time of transplantation, laparotomy including tumor staging will be performed and if there is no sign of extrahepatic disease, liver transplantation will continue according to institutional protocols. Participants will be followed for 5 years and monitored for safety, survival and disease recurrence.

Regarding the translational research:

* The metastatic liver removed on day of transplant will be analysed using high-throughput single-cell RNA sequencing (scRNA-seq) which will allow deep phenotyping of cells for detection of rare and common cell populations and determination of developmental trajectories of distinct cell lineages.
* RAS allele fraction will be monitored by BEAMing and it will be performed before chemotherapy treatment, before LT, post-transplantation, and every 3 months until the patient relapses if relapses.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent.
2. Male or female, aged 18-70 years old inclusive at study entry.
3. ECOG (Eastern Cooperative Oncology Group) 0 or 1.
4. Histologically-proven primary colorectal tumor.
5. Bilateral, limited at liver and non-resectable CRLM by consensus in Multidisciplinary Committee.
6. Resection of primary colorectal tumor according oncological principles and adequate TNM stage.
7. Time from primary colorectal tumor resection to transplant ≥ 12 months.
8. Primary colorectal tumor stage ≤ T3N1. If time between primary tumor resection is ≥ 2 years, stage T4N0 or T4N2 is accepted.
9. No signs of extrahepatic metastatic disease according to PET/CT scan, CT and pelvic MRI.
10. The patient has undergone systemic chemotherapy for a minimum of 3 months at the time of screening and maximum of 2 lines of fluoropyrimidine based chemotherapy combined or not with irinotecan or oxaliplatin associated or no not with targeted therapy based in molecular biomarkers.
11. Demonstrated stability or partial regression of CRLM following RECIST criteria v 1.1., at minimum 3 months since the last treatment received and immediately prior to screening.
12. CEA (Carcinoembryonic antigen) values ≤ 80 µg/L immediately prior to screening.
13. Adequate blood test regarding:

    * Creatinine ≤1.25 x upper normal level or estimated glomerular filtration rate (eGFR) ≥60 mL/min/1.73m2 using following the Chronic Kidney disease epidemiology collaboration (CKD-EPI) formula.
    * Platelets ≥80 × 109/L
    * Neutrophiles ≥ 2.5 × 109/L
14. Patients with hepatic failure after resection will be considered if it occurs as a consequence of an inadequate preoperative estimation of the functional volume that would have contraindicated the surgery. They should meet the inclusion criteria and none of the exclusion criteria.

Exclusion Criteria:

1. Largest Lesion >5.5cm immediately prior to screening
2. Patients with Lynch Syndrome
3. BRAF mutation and/or primary tumor of microsatellite instability (MSI)
4. Recurrence of primary tumor confirmed by colonoscopy or pelvic MRI within the last 12 months prior to screening.
5. Previous or concurrent cancer in the last 5 years. Any cancer curatively treated 5 years prior to entry or treated basal cell carcinoma is permitted.
6. Substance abuse, medical, psychological or social conditions that may interfere with the patient´s participation in the study or evaluation of the study results.
7. Cardiac or pulmonary disease uncontrolled as contraindication for any surgical procedure.
8. Active infection.
9. Pregnant or breast-feeding patients
10. Any reason why in the opinion of the investigator, the patient should not participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Five years overall survival | 5 years
  Percentage of subject who reach the endpoint of overall survival from the inclusion in waiting list until death or last follow-up

SECONDARY OUTCOMES:
One and three years overall survival | 1 and 3 years
  Percentage of subjects who reach the endpoint of overall survival from the inclusion in waiting list until death or last follow-up
One, three and five years recurrence free survival | 1, 3 and 5 years
  Percentage or patients who did not progress from transplantation until death or last follow-up analysed using Kaplan-Meier and the log-rank test.
Number of patients that drop-out of the study prior to receive intervention | Prior to liver transplantation
  Percentage of patients that drop-out of the study prior to liver transplantation
Patterns of cancer recurrence after liver transplantation | 5 years
  Defined as porcentage of patients with hepatic recurrence, extrahepatic recurrence or both
Changes in quality of life assessed by EORTC QLQ-C30 questionnaire (European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30) | 5 years
  These questions allowed categorizing patients into whether they exhibited a clinically important symptom/functional impairment for each scale from 1 (not at all) to 4 (very much). It would be assessed pretransplantation and every 6 months after transplantation.

OTHER OUTCOMES:
Percentage of the intratumoral genetic heterogeneity of the metastatic liver through an in-depth lineage study | On day of transplantation
  High-throughput single-cell RNA sequencing (scRNA-seq) will allow deep phenotyping of cells, allowing detection of rare and common cell populations and determination of developmental trajectories of distinct cell lineages from the metastatic liver removed to the recurrence (hepatic or extrahepatic).
Percentage of patients with circulating tumor DNA (ctDNA) | 5 years
  ctDNA monitorization will be performed pre-chemotherapy, pre-transplantation and every three months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Charco, Principal Investigator — Department of HPB Surgery and Transplants, Hospital Universitario Vall d´Hebron; Elena Elez, Principal Investigator — Department of Oncology, Hospital Universitario Vall d´Hebron; Cristina Dopazo, Principal Investigator — Department of HPB Surgery and Transplants, Hospital Universitario Vall d´Hebron; Ernest Hidalgo, Study Chair — Department of HPB Surgery and Transplants, Hospital Universitario Vall d´Hebron; Itxarone Bilbao, Study Chair — Department of HPB Surgery and Transplants, Hospital Universitario Vall d´Hebron; Concepción Gómez-Gavara, Study Chair — Department of HPB Surgery and Transplants, Hospital Universitario Vall d´Hebron; Mireia Caralt, Study Chair — Department of HPB Surgery and Transplants, Hospital Universitario Vall d´Hebron; Javier Ros, Study Chair — Department of Oncology, Hospital Universitario Vall d´Hebron; Francesc Salva, Study Chair — Department of Oncology, Hospital Universitario Vall d´Hebron; Isabel Campos-Varela, Study Chair — Liver Unit, Department of Internal Medicine, Hospital Universitario Vall d´Hebron; Lluis Castells, Study Chair — Liver Unit, Department of Internal Medicine, Hospital Universitario Vall d´Hebron
Locations (1):
- Department of HPB Surgery and Transplants, Hospital Vall d´Hebron, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reinert T, Henriksen TV, Christensen E, Sharma S, Salari R, Sethi H, Knudsen M, Nordentoft I, Wu HT, Tin AS, Heilskov Rasmussen M, Vang S, Shchegrova S, Frydendahl Boll Johansen A, Srinivasan R, Assaf Z, Balcioglu M, Olson A, Dashner S, Hafez D, Navarro S, Goel S, Rabinowitz M, Billings P, Sigurjonsson S, Dyrskjot L, Swenerton R, Aleshin A, Laurberg S, Husted Madsen A, Kannerup AS, Stribolt K, Palmelund Krag S, Iversen LH, Gotschalck Sunesen K, Lin CJ, Zimmermann BG, Lindbjerg Andersen C. Analysis of Plasma Cell-Free DNA by Ultradeep Sequencing in Patients With Stages I to III Colorectal Cancer. JAMA Oncol. 2019 Aug 1;5(8):1124-1131. doi: 10.1001/jamaoncol.2019.0528. PMID 31070691
- [Background] Elez E, Chianese C, Sanz-Garcia E, Martinelli E, Noguerido A, Mancuso FM, Caratu G, Matito J, Grasselli J, Cardone C, Esposito Abate R, Martini G, Santos C, Macarulla T, Argiles G, Capdevila J, Garcia A, Mulet N, Maiello E, Normanno N, Jones F, Tabernero J, Ciardello F, Salazar R, Vivancos A. Impact of circulating tumor DNA mutant allele fraction on prognosis in RAS-mutant metastatic colorectal cancer. Mol Oncol. 2019 Sep;13(9):1827-1835. doi: 10.1002/1878-0261.12547. Epub 2019 Jul 31. PMID 31322322
- [Background] Dueland S, Grut H, Syversveen T, Hagness M, Line PD. Selection criteria related to long-term survival following liver transplantation for colorectal liver metastasis. Am J Transplant. 2020 Feb;20(2):530-537. doi: 10.1111/ajt.15682. Epub 2019 Nov 28. PMID 31674105
- [Background] Bonney GK, Chew CA, Lodge P, Hubbard J, Halazun KJ, Trunecka P, Muiesan P, Mirza DF, Isaac J, Laing RW, Iyer SG, Chee CE, Yong WP, Muthiah MD, Panaro F, Sanabria J, Grothey A, Moodley K, Chau I, Chan ACY, Wang CC, Menon K, Sapisochin G, Hagness M, Dueland S, Line PD, Adam R. Liver transplantation for non-resectable colorectal liver metastases: the International Hepato-Pancreato-Biliary Association consensus guidelines. Lancet Gastroenterol Hepatol. 2021 Nov;6(11):933-946. doi: 10.1016/S2468-1253(21)00219-3. Epub 2021 Sep 8. PMID 34506756